CLINICAL TRIAL: NCT02685761
Title: Randomized Controlled Trial of Wound Complication Rates Between Low Transverse, Midline Vertical, and High Transverse Skin Incisions in Women With a BMI of 40 or Above Undergoing a Cesarean Section for Delivery
Brief Title: Skin Incisions and Wound Complication Rates for C-sections in Obese Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Peter R Cole, MD, Chief, Divison of Gynecology, Department of OBGYN, Albany Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4128
Record Dates: First submitted 2016-02-16; First posted 2016-02-19 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Obesity; Infection; Cesarean Section; Surgical Wound
MeSH Terms: conditions — Obesity; Infections; Surgical Wound

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low Transverse (No Intervention): Patients in this arm will undergo their cesarean section using the standard low transverse skin incision location
- Midline Vertical (Experimental): Patients in this arm will undergo their cesarean section using a midline vertical skin incision
  Interventions: Procedure: Midline Vertical
- High Transverse (Experimental): Patients in this arm will undergo their cesarean section using a high transverse skin incision, above the pannus
  Interventions: Procedure: High Transverse

INTERVENTIONS:
Procedure: Midline Vertical — Cesarean section performed using a midline vertical skin incision, located between the umbilicus and pubis
  Arms: Midline Vertical
Procedure: High Transverse — Cesarean section performed using a transverse skin incision located above the pannus
  Arms: High Transverse

SUMMARY:
It is the purpose of this study to evaluate the relationship between a low transverse, vertical midline, and supra-panicular high transverse skin incisions and the rate of wound complications in women with a BMI of 40 or greater undergoing a cesarean section for delivery. So far, the choice of incision for the morbidly obese is based only on case reports. No randomized controlled trials have been done up to date comparing these methods. It is our hope that a high transverse incision will have all of the benefits of a low transverse skin incision, with the added benefit of better exposure offered by a vertical midline incision, without the added increased risk of subjecting the woman to a vertical hysterotomy.

ELIGIBILITY:
Inclusion Criteria:

* pre-pregnancy BMI equal or greater than 40

Exclusion Criteria:

* prior cesarean section or laparotomy

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 309 (Estimated)
Dates: Start 2015-09; Primary Completion 2020-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Wound Complications | 6 months

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Albany Medical Center Obstetrics and Gynecology, Albany, New York
  - Albany Medical Center, Albany, New York
  - Albany Medical Center Obstetrics and Gynecology, Ballston Spa, New York
  - Albany Medical Center Obstetrics and Gynecology, Clifton Park, New York
  - Albany Medical Center Obstetrics and Gynecology, Delmar, New York
  - Albany Medical Center Obstetrics and Gynecology, Latham, New York

IPD SHARING:
Plan to Share IPD: No